CLINICAL TRIAL: NCT03393975
Title: A Phase 3, Prospective, Randomized, Controlled, Open-label, Multicenter, 2 Period Crossover Study With a Single Arm Continuation Evaluating the Safety And Efficacy of BAX 930 (rADAMTS13) in the Prophylactic And On-demand Treatment of Subjects With Severe Congenital Thrombotic Thrombocytopenic Purpura (cTTP, Upshaw-Schulman Syndrome [USS], Hereditary Thrombotic Thrombocytopenic Purpura [hTTP])
Brief Title: A Study of BAX 930 in Children, Teenagers, and Adults Born With Thrombotic Thrombocytopenic Purpura (TTP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 281102; 2017-000858-18 (EudraCT Number); TAK-755-281102 (Other: Sponsor)
Record Dates: First submitted 2017-10-05; First posted 2018-01-09 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — ADAMTS13 protein, human; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, prospective, randomized, controlled, open-label, multicenter, 2-period crossover study with a single arm continuation evaluating the safety and efficacy of BAX 930 in the prophylactic and on-demand treatment of participants with severe congenital thrombotic thrombocytopenic purpura (cTTP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Prophylaxis Cohort I: TAK-755 Then SoC (Experimental): Participants received a single intravenous (IV) infusion of 40 international units per kilogram (IU/kg) rADAMTS13 manufactured in Orth, Austria (TAK-755 ORT), every 2 weeks (Q2W) for 6 months in Period 1 followed by standard of care (SoC) for 6 months in Period 2. Thereafter participants received rADAMTS13 manufactured in Singapore (TAK-755 SIN), dose IV infusion of 40 IU/kg Q2W for 6 months in Period 3. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
  Interventions: Biological: TAK-755; Biological: Standard of care
- Prophylaxis Cohort II: SoC Then TAK-755 (Experimental): Participants received SoC for 6 months in Period 1 followed by IV infusions of 40 IU/kg dose of TAK-755 ORT Q2W in Period 2 for the next 6 months. Thereafter participants received TAK-755 SIN dose IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
  Interventions: Biological: TAK-755; Biological: Standard of care
- On Demand Cohort I: TAK-755 (Experimental): Participants experiencing an acute TTP event who met all other inclusion criteria and entered the study through the TAK-755 cohort of the Urgent Treatment Period received initial dose of IV infusion 40 IU/kg [+/- 4 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 1 followed by a subsequent dose IV infusions of 20 IU/kg [+/- 2 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 2 and an additional daily dose IV infusions of 15 IU/kg [+/- 1.5 IU/kg] TAK-755 on Day 3 until 2 days after the acute event was resolved. Upon resolution of the acute TTP event, participants had the option to either move to the prophylaxis cohort of the study or discontinue entirely.
  Interventions: Biological: TAK-755
- On Demand Cohort II: SoC (Experimental): Participants experiencing an acute TTP event who met all other inclusion criteria and entered the study through the SoC cohort of the Urgent Treatment Period received the investigator-recommended SoC and dosing regimen until the acute event was resolved. Upon resolution of the acute TTP event, participants had the option to either move to the prophylaxis cohort of the study or discontinue entirely.
  Interventions: Biological: Standard of care

INTERVENTIONS:
Biological: TAK-755 — Participants in prophylaxis cohort will receive IV infusions of 40 IU/kg TAK-755 ORT during Period 1 and Period 2 and switch to TAK-755 SIN during Period 3 for six months once in a week or twice in a week. In On-demand cohort participants will receive daily IV dose of TAK-755.
  Other Names: rADAMTS13; SHP-655; recombinant ADAMTS13; BAX 930
  Arms: On Demand Cohort I: TAK-755; Prophylaxis Cohort I: TAK-755 Then SoC; Prophylaxis Cohort II: SoC Then TAK-755
Biological: Standard of care — Participants will receive Investigator-recommended Standard of care (SoC).
  Arms: On Demand Cohort II: SoC; Prophylaxis Cohort I: TAK-755 Then SoC; Prophylaxis Cohort II: SoC Then TAK-755

SUMMARY:
Thrombotic thrombocytopenic purpura (or TTP for short) is a condition where blood clots form in small blood vessels throughout the body. The clots can limit or block the flow of oxygen-rich blood to the body's organs, such as the brain, kidneys, and heart. As a result, serious health problems can develop. The increased clotting that occurs in TTP uses up the cells that help the blood to clot, called platelets. With fewer platelets available in the blood, bleeding problems can occur. People who have TTP may bleed underneath the skin forming purple bruises or purpura, or from the surface of the skin. TTP also can cause anemia, a condition in which red blood cells break apart faster than the body can replace them leading to lower than normal number of red blood cells.

A lack of activity in the ADAMTS13 enzyme, a protein in the blood involved in blood clotting, causes TTP. The enzyme breaks up another blood protein called von Willebrand factor that clumps together with platelets to form blood clots. Some people are born with this condition, others get the condition during their life. Many people who born with TTP experience frequent flareups that need to be treated right away. If not treated It can be fatal or cause lasting damage, such as brain damage or a stroke. BAX 930 is a medicine that replaces ADAMTS13 and can prevent or control TTP flareups, called TTP events.

The main aim of this study is to compare the number of TTP events in people born with severe TTP when they treated with BAX 930 versus when they are treated with the standard treatment. Treatment will be given in 2 ways:

* BAX 930 or standard treatment given to prevent TTP events from happening.
* BAX 930 or standard treatment given to control an acute TTP event when it happens, according to the clinic's standard practice.

Both BAX 930 and standard treatment are given slowly through a vein (infusion).

At the first visit, the study doctor will check if you can participate in the study. If you are eligible and enter the study, you will follow an assigned schedule and either start with BAX 930 (Period 1) and then switch to standard treatment (Period 2) or start with standard treatment (Period 1) and then switch to BAX 930 (Period 2). Everyone will be treated with BAX 930 again for Period 3. Each Period will last approximately 6 months.

If you enter the study to control an acute TTP event, you will follow a schedule receiving either BAX 930 or standard care to treat your acute TTP event. Once the acute TTP event has gotten better, you can decide to continue in the study and be given treatment to prevent TTP events from happening, following the schedule above.

Another study's aim is to assess side effects from treatment with BAX 930 and standard treatment. To do that, the study doctor will ask you questions about your health at each study visit.

The study doctors will also check how long BAX 930 stays in the blood of the participants, over time. They will do this from blood samples taken after participants receive their specific infusions of BAX 930. This will happen at different times during the study.

1 month after all treatment has been completed, participants will visit the clinic for a final check-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative has provided signed informed consent >= 18 years of age and/or assent form (signed by legal representative if participants is <18 years of age).
* Participant is 0 to 70 years of age, inclusive, at the time of screening. (Participants < 18 years of age will be enrolled only after at least 5 adults (>= 18 years of age) each have at least 10 exposures with BAX 930 and reviewed by the Data Monitoring Committee (DMC). In France, no participants younger than 18 years of age will be enrolled into the study before the first adult participant has been treated with BAX 930 for a minimum of 6 months.
* Participant has a documented diagnosis of severe hereditary ADAMTS13 deficiency, defined as:

  * Confirmed by molecular genetic testing, documented in participant history or at screening, and
  * ADAMTS13 activity < 10 % as measured by the fluorescent resonance energy transfer- von Willebrand factor73 (FRETS-VWF73) assay, documented in participant history or at screening (participants currently receiving standard of care (SoC) prophylactic therapy may exceed 10% ADAMTS13 activity at screening).

Note: Participants currently receiving prophylactic therapy will be screened immediately prior to their usual prophylactic infusion

* Participant does not display any severe thrombotic thrombocytopenic purpura (TTP) signs (platelet count < 100,000/ microliter (mcL) and elevation of lactate dehydrogenase (LDH) greater than (>2)* ULN) at screening. (Prophylactic cohort only).
* Participant is currently on a prophylactic dosing regimen or has a documented history of at least 1 TTP event and an ability to tolerate SoC prophylactic dosing (prophylactic cohort only).
* Participants >= 16 years of age must have a Karnofsky score >= 70% and participants < 16 years of age must have a Lansky score >= 80%.
* Participant is hepatitis C virus (HCV)-negative as confirmed by antibody or polymerase chain reaction testing OR HCV-positive if their disease is chronic but stable.
* If female of childbearing potential, participant presents with a negative blood or urine pregnancy test, confirmed no more than 7 days before the first administration, and agrees to employ adequate birth control measures for the duration of the study and to undergo quarterly pregnancy testing.
* Sexually active males must use an accepted and effective method of contraception during the treatment and until a minimum of 16 days after the last dose administered.
* Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Participant has been diagnosed with any other TTP-like disorder (microangiopathic hemolytic anemia), including acquired TTP.
* Participant has known hypersensitivity to hamster proteins.
* Participant has experienced an acute TTP event less than 30 days prior to screening (prophylactic cohort only).
* Participant has a medical history or presence of a functional ADAMTS13 inhibitor at screening.
* Participant has a medical history of genetic or acquired immune deficiency that would interfere with the assessment of product immunogenicity, including participants who are human immunodeficiency virus (HIV)-positive with an absolute cluster of differentiation 4 (CD4) count < 200/ cubic millimeter (mm^3) or who are receiving chronic immunosuppressive drugs.
* Participant has been diagnosed with severe cardiovascular disease (New York Heart Association classes 3 to 4).
* Participant with end stage renal disease requiring chronic dialysis.
* Participant has been diagnosed with hepatic dysfunction, as evidenced by, but not limited to, any of the following:

  * Serum alanine aminotransferase (ALT) >= 2* ULN.
  * Severe hypoalbuminemia < 24 gram per liter (g/L).
  * Portal vein hypertension (e.g., presence of otherwise unexplained splenomegaly, history of esophageal varices).
* In the opinion of the investigator, the participant has another clinically significant concomitant disease that may pose additional risks for the participant.
* Participant has been treated with an immunomodulatory drug, excluding topical treatment (e.g., ointments, nasal sprays), within 30 days prior to enrollment. Use of corticosteroids in conjunction with administration of fresh frozen plasma (FFP) to prevent allergic reactions is permitted.
* Participant has an acute illness (e.g., influenza, flu-like syndrome, allergic rhinitis/conjunctivitis, bronchial asthma) at the time of screening (prophylaxis cohort only).
* Participant is receiving or anticipates receiving another investigational drug and/or interventional drug within 30 days before enrollment.
* Participant has a history of drug and/or alcohol abuse within the last 2 years.
* Participant has a progressive fatal disease and/or life expectancy of less than 3 months.
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
* Participant suffers from a mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude.
* Participant is a family member or employee of the sponsor or investigator.
* If female, participant is pregnant or lactating at the time of enrollment.
* Any contraindication to SoC medicinal product(s) as per local prescribing information.

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (33):
- United States (7):
  - Winship Cancer Institute, Atlanta, Georgia
  - Alliance for Childhood Diseases, Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State Univ College Of Medicine, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - The Methodist Hospital, Houston, Texas
- AKH - Medizinische Universität Wien, Vienna, Austria
- France (5):
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hôpital Necker - Enfants Malades, Paris, Paris
  - Hôpital Saint-Antoine, Paris, Paris
  - CHU Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez Cedex, Pays de la Loire Region
  - Hôpital Robert Debré - Paris, Paris
- Germany (2):
  - Universitaetsklinikum Jena, Jena, Thuringia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliera Universitaria "Policlinico - Vittorio Emanuele" (Presidio Ferrarotto Alessi), Catania
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Dipartimento di Medicina Traslazionale e di Precisione - "Sapienza" Universita di Roma, Rome
- Japan (3):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City, Tokyo-To
- Poland (2):
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - University College London Hospitals, London, Greater London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Scully M, Antun A, Cataland SR, Coppo P, Dossier C, Biebuyck N, Hassenpflug WA, Kentouche K, Knobl P, Kremer Hovinga JA, Lopez-Fernandez MF, Matsumoto M, Ortel TL, Windyga J, Bhattacharya I, Cronin M, Li H, Mellgard B, Patel M, Patwari P, Xiao S, Zhang P, Wang LT; cTTP Phase 3 Study Investigators. Recombinant ADAMTS13 in Congenital Thrombotic Thrombocytopenic Purpura. N Engl J Med. 2024 May 2;390(17):1584-1596. doi: 10.1056/NEJMoa2314793. PMID 38692292
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc84db2bf003ab4602d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 13 October 2017 to 30 May 2024.
Pre-assignment Details: Participants with a diagnosis of severe congenital thrombotic thrombocytopenic purpura (cTTP) were enrolled in either prophylaxis or on demand cohorts. All participants received intravenous infusion of TAK-755 or standard treatment in Prophylaxis Periods 1 and 2, and TAK-755 in Prophylaxis Period 3 (hereafter Prophylaxis Periods 1, 2, and 3 are referred to simply as Periods 1, 2, and 3). 52 participants enrolled into the study but one participant withdrew before being randomized to treatment.
Period: Urgent Treatment Period
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755 | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Started | 0 | 0 | 2 | 4
Safety Analysis Set (The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization and reported as per actual treatment received.) | 0 | 0 | 2 | 4
Full Analysis Set (The Full Analysis Set included all participants with a confirmed cTTP diagnosis who received at least 1 dose of BAX 930 or SoC treatment after randomization.) | 0 | 0 | 2 | 4
Modified Full Analysis Set (Modified Full Analysis Set included all Full Analysis Set participants who were treated according to their randomized treatment sequence with the exclusion of those enrolled prior to November 2017 who were treated with SoC instead of the randomized treatment of TAK-755 in period 1 because TAK-755 was not available. For participants enrolled prior to November 2017, only the first 6 months of SoC treatment in period 1 was included in the analysis.) | 0 | 0 | 2 | 4
Completed | 0 | 0 | 2 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Period: Prophylaxis Period 1
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755 | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Started | 23 | 25 (Only 3 participants from On Demand Cohort II: SoC switched to Prophylactic Cohort II: SoC Then TAK-755.) | 0 | 0
Safety Analysis Set (The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization and reported as per actual treatment received.) | 23 | 25 | 0 | 0
Full Analysis Set (The Full Analysis Set included all participants with a confirmed cTTP diagnosis who received at least 1 dose of BAX 930 or SoC treatment after randomization.) | 23 | 24 | 0 | 0
Modified Full Analysis Set (Modified Full Analysis Set included all Full Analysis Set participants who were treated according to their randomized treatment sequence with the exclusion of those enrolled prior to November 2017 who were treated with SoC instead of the randomized treatment of TAK-755 in period 1 because TAK-755 was not available. For participants enrolled prior to November 2017, only the first 6 months of SoC treatment in period 1 was included in the analysis.) | 21 | 24 | 0 | 0
Completed | 23 | 24 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 0 | 0
Period: Prophylaxis Period 2
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755 | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Started | 23 | 24 | 0 | 0
Completed | 23 | 23 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 0 | 0
Period: Prophylaxis Period 3
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755 | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Started | 23 | 23 | 0 | 0
Completed | 23 | 23 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization. Two participants randomized to Prophylaxis Cohort I received actual treatment as per Prophylaxis Cohort II and are presented per actual treatment arm.
Groups:
- Prophylaxis Cohort I: TAK-755 Then SoC: Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in Period 1 followed by SoC for 6 months in Period 2. Thereafter participants received TAK-755 SIN dose IV infusion of 40 IU/kg Q2W for 6 months in Period 3. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
- On Demand Cohort I: TAK-755: Participants experiencing an acute TTP event who met all other inclusion criteria and entered the study through the TAK-755 cohort of the Urgent Treatment Period received initial dose of IV infusions 40 IU/kg [+/- 4 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 1 followed by a subsequent dose IV infusion of 20 IU/kg [+/- 2 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 2 and an additional daily dose IV infusions of 15 IU/kg [+/- 1.5 IU/kg] TAK-755 on Day 3 until 2 days after the acute event was resolved. Upon resolution of the acute TTP event, participants had the option to either move to the prophylaxis cohort of the study or discontinue entirely.
- Total: Total of all reporting groups
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755 | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC | Total
Number analyzed (Participants) | 21 | 27 | 2 | 4 | 54
Age, Customized [Count of Participants; unit: Participants] — Population: A cohort-wise data representation is used and number analyzed denotes the number of participants in each cohort presented row-wise.
  Participants
    Prophylaxis Cohort: number analyzed (Participants) | 21 | 27 | 0 | 0 | 48
    Prophylaxis Cohort: ≥18 years | 16 | 20 | 0 | 0 | 36
    Prophylaxis Cohort: 12 to <18 years | 1 | 3 | 0 | 0 | 4
    Prophylaxis Cohort: 6 to <12 years | 1 | 3 | 0 | 0 | 4
    Prophylaxis Cohort: <6 years | 3 | 1 | 0 | 0 | 4
    On Demand Cohort: number analyzed (Participants) | 0 | 0 | 2 | 4 | 6
    On Demand Cohort: ≥18 years | 0 | 0 | 2 | 3 | 5
    On Demand Cohort: 12 to <18 years | 0 | 0 | 0 | 0 | 0
    On Demand Cohort: 6 to <12 years | 0 | 0 | 0 | 0 | 0
    On Demand Cohort: <6 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A cohort-wise data representation is used and number analyzed denotes the number of participants in each cohort presented row-wise.
  Participants
    Prophylaxis Cohort: number analyzed (Participants) | 21 | 27 | 0 | 0 | 48
    Prophylaxis Cohort: Female | 12 | 16 | 0 | 0 | 28
    Prophylaxis Cohort: Male | 9 | 11 | 0 | 0 | 20
    On Demand Cohort: number analyzed (Participants) | 0 | 0 | 2 | 4 | 6
    On Demand Cohort: Female | 0 | 0 | 1 | 1 | 2
    On Demand Cohort: Male | 0 | 0 | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A cohort-wise data representation is used and number analyzed denotes the number of participants in each cohort presented row-wise.
  Participants
    Prophylaxis Cohort: number analyzed (Participants) | 21 | 27 | 0 | 0 | 48
    Prophylaxis Cohort: Hispanic or Latino | 1 | 0 | 0 | 0 | 1
    Prophylaxis Cohort: Not Hispanic or Latino | 16 | 23 | 0 | 0 | 39
    Prophylaxis Cohort: Unknown or Not Reported | 4 | 4 | 0 | 0 | 8
    On Demand Cohort: number analyzed (Participants) | 0 | 0 | 2 | 4 | 6
    On Demand Cohort: Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    On Demand Cohort: Not Hispanic or Latino | 0 | 0 | 2 | 4 | 6
    On Demand Cohort: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A cohort-wise data representation is used and number analyzed denotes the number of participants in each cohort presented row-wise.
  Participants
    Prophylaxis Cohort: number analyzed (Participants) | 21 | 27 | 0 | 0 | 48
    Prophylaxis Cohort: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Prophylaxis Cohort: Asian | 2 | 3 | 0 | 0 | 5
    Prophylaxis Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Prophylaxis Cohort: Black or African American | 0 | 1 | 0 | 0 | 1
    Prophylaxis Cohort: White | 15 | 17 | 0 | 0 | 32
    Prophylaxis Cohort: More than one race | 0 | 1 | 0 | 0 | 1
    Prophylaxis Cohort: Unknown or Not Reported | 4 | 5 | 0 | 0 | 9
    On Demand Cohort: number analyzed (Participants) | 0 | 0 | 2 | 4 | 6
    On Demand Cohort: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    On Demand Cohort: Asian | 0 | 0 | 1 | 0 | 1
    On Demand Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    On Demand Cohort: Black or African American | 0 | 0 | 0 | 1 | 1
    On Demand Cohort: White | 0 | 0 | 1 | 2 | 3
    On Demand Cohort: More than one race | 0 | 0 | 0 | 1 | 1
    On Demand Cohort: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Thrombotic Thrombocytopenic Purpura (TTP) Events During Prophylactic Treatment
Description: As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 74.5 months
Population: Modified Full Analysis Set(mFAS): all FAS participants who were treated according to their randomized treatment sequence with exclusion of those enrolled prior to Nov. 2017 who were treated with SoC instead of randomized treatment of TAK-755 in period 1 because TAK-755 was unavailable.For participants enrolled prior to Nov 2017,only first 6 months of SoC treatment in period 1 was included in analysis.Overall number of participants analyzed:number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Prophylaxis Cohort: TAK-755 (Periods 1 and 2): Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in either Period 1 or Period 2. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
- Prophylaxis Cohort: TAK-755 (Period 3): Participants received TAK-755 SIN dose of IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
- Prophylaxis Cohort: SoC (Periods 1 and 2): Participants received SoC for 6 months in either Period 1 or Period 2.
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 0 | 0 | 1

2. Secondary Outcome: Percentage of Acute Thrombotic Thrombocytopenic Purpura (TTP) Events Responding to TAK-755
Description: Percentage of acute TTP events responding to TAK-755, was defined as not requiring the use of another human disintegrin and metalloprotease with a thrombospondin type 1 motif, member 13 (ADAMTS13)-containing agent. As per planned analysis, data for this outcome measure were collected and reported only for the TAK-755 treatment arm of both the prophylaxis (irrespective of the prophylaxis periods) and on demand cohorts.
Time Frame: Up to 79.6 months
Population: mFAS:all FAS participants who were treated according to their randomized treatment sequence with exclusion of those enrolled prior to Nov.2017 who were treated with SoC instead of randomized treatment of TAK-755 in period 1 as TAK-755 was unavailable. For participants enrolled prior to Nov 2017,only first 6 months of SoC treatment in period 1 was included in analysis.Overall number of participants: participants with acute TTP events that were confirmed by central lab data treated with TAK-755.
Measure: Number; unit: percentage of events
Groups:
- Prophylaxis Cohort: TAK-755: Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in either Period 1 or Period 2. Thereafter participants received TAK-755 SIN dose of IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 ORT could be replaced with TAK-755 SIN and vice versa depending on availability and other criteria.
- On Demand Cohort I: TAK-755: Participants experiencing an acute TTP event who met all other inclusion criteria and entered the study through the TAK-755 cohort of the Urgent Treatment Period received initial dose of IV infusions 40 IU/kg [+/- 4 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 1 followed by a subsequent dose IV infusions of 20 IU/kg [+/- 2 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 2 and an additional daily dose IV infusions of 15 IU/kg [+/- 1.5 IU/kg] TAK-755 on Day 3 until 2 days after the acute event was resolved. Upon resolution of the acute TTP event, participants had the option to either move to the prophylaxis cohort of the study or discontinue entirely.
Arm/Group | Prophylaxis Cohort: TAK-755 | On Demand Cohort I: TAK-755
Number analyzed (Participants) | 0 | 1
percentage of events |  | 100

3. Secondary Outcome: Time to Resolution of Acute TTP Events
Description: Time to resolution of acute TTP events following initiation of treatment with TAK-755 or SoC agent was assessed. Acute TPP events were considered resolved when: (a) Platelet count was >150,000 per microliter (μL) or drop of platelet count was within 25 percent (%) of baseline, whichever occurred first, and (b) Elevation of lactate dehydrogenase (LDH) <1.5 x baseline or <1.5 x upper limit of normal (ULN). As per planned analysis, data for this outcome measure were collected and reported in a combined manner irrespective of the prophylaxis treatment Periods, partitioned per treatment received (TAK-755 and SoC) for the on demand and prophylactic cohorts.
Time Frame: Up to 79.6 months
Population: mFAS: all FAS participants who were treated according to their randomized treatment sequence with exclusion of those enrolled prior to Nov. 2017 who were treated with SoC instead of randomized treatment of TAK-755 in period 1 as TAK-755 was unavailable. For participants enrolled prior to Nov. 2017,only first 6 months of SoC treatment in period 1 was included in analysis.Overall number of participants analyzed:number of participants with acute TTP events that were confirmed by central lab data.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Prophylaxis Cohort: SoC: Participants received SoC for 6 months in either Period 1 or Period 2.
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 0 | 1 | 1 | 1
days |  | 14.8 [NA to NA] — 95% confidence interval was not estimable due to censoring. | 3.0 [NA to NA] — 95% confidence interval was not estimable due to censoring. | 1.5 [NA to NA] — 95% confidence interval was not estimable due to censoring.

4. Secondary Outcome: Number of Participants With Thrombocytopenia During Prophylactic Treatment
Description: Thrombocytopenia was defined as a decrease in platelet count ≥25 % of baseline or a platelet count <150,000/μL, reported by treatment arm for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: mFAS included all FAS participants who were treated according to their randomized treatment sequence with exclusion of those enrolled prior to Nov. 2017 who were treated with SoC instead of randomized treatment of TAK-755 in period 1 as TAK-755 was unavailable. For participants enrolled prior to Nov. 2017, only first 6 months of SoC treatment in period 1 was included in analysis. Overall number of participants analyzed indicates the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 13 | 11 | 21

5. Secondary Outcome: Number of Participants With Microangiopathic Hemolytic Anemia During Prophylactic Treatment
Description: Microangiopathic hemolytic anemia was defined as an elevation of LDH >1.5* of baseline or >1.5*ULN (with a possible evidence of schistocytes on blood smear) and was reported by treatment arm for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 8 | 13 | 12

6. Secondary Outcome: Number of Participants With Neurological Symptoms During Prophylactic Treatment
Description: Neurological symptoms (TTP related) (e.g., confusion, dysphonia, dysarthria, focal or general motor symptoms including seizures), were reported by treatment arm for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 4 | 9 | 7

7. Secondary Outcome: Number of Participants With Renal Dysfunction During Prophylactic Treatment
Description: Renal dysfunction was defined as an increase in serum creatinine >1.5*baseline. Number of participants with renal dysfunction were reported by treatment arm for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 5 | 4 | 2

8. Secondary Outcome: Number of Participants With Abdominal Pain During Prophylactic Treatment
Description: Number of participants with abdominal pain (TTP related) were reported by treatment arm for the prophylaxis cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 2 | 2 | 6

9. Secondary Outcome: Number of Supplemental Doses Prompted by Subacute TTP Event During Prophylactic Treatment
Description: Number of supplemental doses prompted by subacute TTP events were reported by treatment for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Number; unit: supplemental doses
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
supplemental doses | 0 | 5 | 9

10. Secondary Outcome: Number of Participants With Dose Modification Not Prompted by an Acute TTP Event During Prophylactic Treatment
Description: Number of participants with dose modification not prompted by an acute TTP event were reported by treatment for the prophylactic cohort. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 0 | 1 | 3

11. Secondary Outcome: Number of Participants With Acute TTP Events on Their Final Dose
Description: Number of participants with acute TTP events on their final dose and dosing regimen for the prophylactic cohort were reported. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts, in a combined manner for Periods 1 and 2 for TAK-755 and SoC treatments respectively, and separately for Period 3 in which all participants received TAK-755.
Time Frame: Up to 79.6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 (Periods 1 and 2) | Prophylaxis Cohort: TAK-755 (Period 3) | Prophylaxis Cohort: SoC (Periods 1 and 2)
Number analyzed (Participants) | 44 | 44 | 45
Participants | 0 | 0 | 1

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Treatment Emergent Adverse Events (Serious TEAEs)
Description: AE: Any untoward medical occurrence in participants administered IP that does not necessarily have a causal relationship with treatment. TEAE: AE that has start date-time on/after start date-time of first dose of treatment participant is taking on that assessment/period or if it has start date-time before start date-time of first dose but increases in severity on/after start date-time of the first dose of treatment. SAE: An untoward medical occurrence that at any dose meets 1 or more of following criteria: death; initial/prolonged in-patient hospitalization; life threatening experience; persistent/significant disability/incapacity; congenital anomaly, medically important event (may not be immediately life threatening or result in death or require hospitalization but may require medical or surgical intervention to prevent 1 of the other outcomes). Vital signs, clinical chemistry, hematology as assessed by the investigator were reported as AE.
Time Frame: Up to 79.6 months
Population: The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization. As per planned analysis, data for this outcome measure were collected and reported in a combined manner irrespective of the Prophylaxis Periods and partitioned as per the treatment received during the course of the study, presented for the on demand and prophylaxis cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 47 | 48 | 2 | 4
Participants
  TEAES | 42 | 44 | 0 | 3
  Serious TEAEs | 6 | 8 | 0 | 1

13. Secondary Outcome: Number of Participants With Inhibitory Antibodies to ADAMTS13
Description: Number of participants with inhibitory antibodies to ADAMTS13 were reported. As per planned analysis, data for this outcome measure were collected and reported in a combined manner irrespective of the Prophylaxis Periods and partitioned as per the treatment received during the course of the study, presented for the prophylaxis cohorts only.
Time Frame: Up to 79.6 months
Population: The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization. Overall number of participants analyzed is the number of participants with at least one assessment of the targeted parameter in the specified treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 6 | 4
Participants | 1 | 0

14. Secondary Outcome: Total Quantity of ADAMTS13 Administered During the Treatment of Acute TTP Events in Participants in TAK-755 Treatment Arm
Description: Total quantity of ADAMTS13 administered during the treatment of acute TTP events (all acute TTP events irrespective of central lab confirmation were included) was assessed. Acute TTP events typically require 3 to 4 days of intensified treatment. As per planned analysis, data for this outcome measure were collected and reported only for the TAK-755 treatment arm of both the prophylaxis (irrespective of the prophylaxis periods) and on demand cohorts.
Time Frame: Up to 79.6 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Prophylaxis Cohort: TAK-755 | On Demand Cohort I: TAK-755
Number analyzed (Participants) | 0 | 2
IU |  | 5720.25 (189.858)

15. Secondary Outcome: Incremental Recovery (IR) of ADAMTS13 Activity for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: ADAMTS13 activity was measured by the fluorescent resonance energy transfer (FRETS) assay. IR was defined as body weight normalized maximum increase in plasma ADAMTS13 activity level. IR of ADAMTS13 activity for SoC agent and TAK-755 in plasma was assessed. (IU/mL)/(IU/kg) stands for (International units per milliliter)/(International units per kilogram). PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1, end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: PK-I (Month 1:Day 1 up to 12), PK-II (Month 12:Day 1 up to 12), and PK-III (Month 19:Day 1 up to 12): Pre-infusion and at multiple timepoints post-infusion up to 288 hours
Population: The PK Analysis Set included all FAS participants who had adequate post-dose PK measurements for at least one of the PK analytes without major protocol deviations or events that may affect the integrity of the PK data. Overall number of participants analyzed indicates the number of participants with data available for analyses. Number analyzed indicates the number of participants with data available for analyses in the specified category.
Measure: Mean (Standard Deviation); unit: (IU/mL)/(IU/kg)
Groups:
- Prophylaxis Cohort: TAK-755 ORT: Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in either Period 1 or Period 2. TAK-755 ORT could also be continued in Period 3 depending on availability of TAK-755 SIN and other criteria.
- Prophylaxis Cohort: TAK-755 SIN: Participants received TAK-755 SIN dose of IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 SIN could also be given in Periods 1 and 2 depending on availability of TAK-755 ORT and other criteria.
- Prophylaxis Cohort: SoC: Participants received SoC for 6 months in either Period 1 or Period 2 (except for PK-II where they did not receive SoC).
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 36 | 22 | 22
(IU/mL)/(IU/kg)
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 36 | 1 | 22
  PK-I: ADAMTS13 Activity | 0.025 (0.00592) | NA (NA) — Mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification. | 0.0212 (0.0267)
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 26 | 22 | 0
  PK-II: ADAMTS13 Activity | 0.0283 (0.00644) | 0.0292 (0.00630) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 15 | 0
  PK-III: ADAMTS13 Activity |  | 0.0260 (0.00617) |

16. Secondary Outcome: IR of ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: ADAMTS13 antigen was measured using a commercial ADAMTS13 enzyme-linked immunosorbent assay (ELISA) employing ADAMTS13 antigen. IR was defined as body weight normalized maximum increase in plasma ADAMTS13 antigen. IR of ADAMTS13 antigen for SoC agent and TAK-755 in plasma was assessed. (µg/mL)/ (µg/kg) stands for (microgram per milliliter)/(microgram per kilogram). PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1, end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: (µg/mL)/ (µg/kg)
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 37 | 24 | 23
(µg/mL)/ (µg/kg)
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 37 | 1 | 23
  PK-I: ADAMTS13 Antigen | 0.0299 (0.00638) | NA (NA) — Mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification. | 0.0186 (0.00605)
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 25 | 24 | 0
  PK-II: ADAMTS13 Antigen | 0.0339 (0.0080) | 0.0324 (0.00668) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 13 | 0
  PK-III: ADAMTS13 Antigen |  | 0.0264 (0.0102) |

17. Secondary Outcome: Area Under the Plasma Curve [AUC]All of ADAMTS13 Activity for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: h*IU/mL denotes for hours*international units per milliliters. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 33 | 22 | 31
h*IU/mL
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 33 | 0 | 31
  PK-I: ADAMTS13 Activity | 44.15 (11.197) |  | 10.56 (8.263)
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 26 | 22 | 0
  PK-II: ADAMTS13 Activity | 52.83 (11.940) | 52.98 (13.358) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 7 | 0
  PK-III: ADAMTS13 Activity |  | 65.65 (23.487) |

18. Secondary Outcome: AUCall of ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: h*µg/mL denotes for hours*microgram per milliliters. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: h*µg/mL
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 34 | 24 | 31
h*µg/mL
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 34 | 0 | 31
  PK-I: ADAMTS13 Antigen | 34.12 (9.646) |  | 7.590 (6.1344)
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 25 | 24 | 0
  PK-II: ADAMTS13 Antigen | 38.79 (8.835) | 38.95 (11.137) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 6 | 0
  PK-III: ADAMTS13 Antigen |  | 49.74 (19.147) |

19. Secondary Outcome: Terminal Half-Life (t1/2) of ADAMTS13 Activity and ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 34 | 24 | 22
hours
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 33 | 0 | 22
  PK-I: ADAMTS13 Activity | 47.14 (11.573) |  | 62.88 (28.927)
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 34 | 0 | 16
  PK-I: ADAMTS13 Antigen | 53.59 (13.354) |  | 58.70 (23.575)
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 26 | 22 | 0
  PK-II: ADAMTS13 Activity | 52.51 (15.579) | 45.77 (10.231) |
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 25 | 24 | 0
  PK-II: ADAMTS13 Antigen | 54.15 (16.553) | 49.72 (15.942) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 7 | 0
  PK-III: ADAMTS13 Activity |  | 35.38 (5.286) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 6 | 0
  PK-III: ADAMTS13 Antigen |  | 39.85 (3.243) |

20. Secondary Outcome: Mean Residence Time Extrapolated to Infinity (MRT0-inf) of ADAMTS13 Activity and ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: as for outcome 19
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Prophylaxis Cohort: TAK-755-ORT: Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in either Period 1 or Period 2. TAK-755 ORT could also be continued in Period 3 depending on availability of TAK-755 SIN and other criteria.
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 31 | 23 | 2
hours
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 31 | 0 | 2
  PK-I: ADAMTS13 Activity | 64.35 (17.498) |  | NA (NA) — The mean and SD were not estimable as the values were below the lower limit of quantification.
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 31 | 0 | 2
  PK-I: ADAMTS13 Antigen | 71.20 (16.538) |  | NA (NA) — The mean and SD were not estimable as the values were below the lower limit of quantification.
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 25 | 21 | 0
  PK-II: ADAMTS13 Activity | 65.89 (13.472) | 61.56 (11.762) |
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 23 | 23 | 0
  PK-II: ADAMTS13 Antigen | 72.36 (19.224) | 66.30 (18.738) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 7 | 0
  PK-III: ADAMTS13 Activity |  | 41.67 (6.171) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 5 | 0
  PK-III: ADAMTS13 Antigen |  | 46.30 (4.266) |

21. Secondary Outcome: Clearance (CL) of ADAMTS13 Activity and ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: as for outcome 19
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 31 | 23 | 2
liters per hour (L/h)
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 31 | 0 | 2
  PK-I: ADAMTS13 Activity | 0.0618 (0.0144) |  | NA (NA) — Mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification.
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 31 | 0 | 1
  PK-I: ADAMTS13 Antigen | 0.0456 (0.0117) |  | NA (NA) — Mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification.
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 25 | 21 | 0
  PK-II: ADAMTS13 Activity | 0.0530 (0.0134) | 0.0549 (0.0117) |
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 23 | 23 | 0
  PK-II: ADAMTS13 Antigen | 0.0409 (0.0109) | 0.0480 (0.0133) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 7 | 0
  PK-III: ADAMTS13 Activity |  | 0.0553 (0.0177) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 5 | 0
  PK-III: ADAMTS13 Antigen |  | 0.0462 (0.0110) |

22. Secondary Outcome: Volume at Steady State (Vss) of ADAMTS13 Activity and ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: as for outcome 19
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Prophylaxis Cohort: TAK-755-ORT: Participants received a single IV infusion of 40 IU/kg TAK-755 ORT Q2W for 6 months in either Period 1 or Period 2..TAK-755 ORT could also be continued in Period 3 depending on availability of TAK-755 SIN and other criteria.
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 31 | 23 | 2
liters
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 31 | 0 | 2
  PK-I: ADAMTS13 Activity | 3.852 (0.916) |  | NA (NA) — The mean and SD were not estimable as the values were below the lower limit of quantification.
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 31 | 0 | 1
  PK-I: ADAMTS13 Antigen | 3.124 (0.650) |  | NA (NA) — The mean and SD were not estimable as the values were below the lower limit of quantification.
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 25 | 21 | 0
  PK-II: ADAMTS13 Activity | 3.401 (0.715) | 3.304 (0.635) |
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 23 | 23 | 0
  PK-II: ADAMTS13 Antigen | 2.812 (0.479) | 3.007 (0.613) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 7 | 0
  PK-III: ADAMTS13 Activity |  | 2.265 (0.669) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 5 | 0
  PK-III: ADAMTS13 Antigen |  | 2.172 (0.698) |

23. Secondary Outcome: Maximum Concentration (Cmax) of ADAMTS13 Activity for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: IU/mL stands for International units per milliliter. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth,Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 36 | 22 | 41
IU/mL
  PK-I: ADAMTS13 Activity: number analyzed (Participants) | 36 | 1 | 41
  PK-I: ADAMTS13 Activity | 1.003 (0.235) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 0.192 (0.102)
  PK-II: ADAMTS13 Activity: number analyzed (Participants) | 26 | 22 | 0
  PK-II: ADAMTS13 Activity | 1.130 (0.253) | 1.162 (0.250) |
  PK-III: ADAMTS13 Activity: number analyzed (Participants) | 0 | 15 | 0
  PK-III: ADAMTS13 Activity |  | 1.036 (0.253) |

24. Secondary Outcome: Cmax of ADAMTS13 Antigen for SoC Agent and TAK-755 in Plasma During Prophylactic Treatment
Description: µg/mL stands for microgram per milliliter. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 37 | 24 | 41
µg/mL
  PK-I: ADAMTS13 Antigen: number analyzed (Participants) | 37 | 1 | 41
  PK-I: ADAMTS13 Antigen | 0.713 (0.145) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 0.141 (0.0710)
  PK-II: ADAMTS13 Antigen: number analyzed (Participants) | 25 | 24 | 0
  PK-II: ADAMTS13 Antigen | 0.804 (0.185) | 0.844 (0.168) |
  PK-III: ADAMTS13 Antigen: number analyzed (Participants) | 0 | 12 | 0
  PK-III: ADAMTS13 Antigen |  | 0.715 (0.203) |

25. Secondary Outcome: Change From Baseline in Assessment of Von Willebrand Factor:Antigen (VWF:Ag) During Prophylactic Treatment
Description: VWF:Ag is a measure of total VWF protein and was assessed using a sandwich ELISA employing polyclonal anti-human-VWF antibodies. Assessments of VWF:Ag at baseline and following infusion of the SoC agent and TAK-755 treatment during the initial PK assessment were reported. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: PK-I (Month 1:Day 12), PK-II (Month 12:Day 12), and PK-III (Month 19:Day 12): Post-infusion at 288 hours
Population: The Pharmacodynamic (PD) Analysis Set included all FAS participants who had at least one valid data point for at least one of the PD outcome measures and had no major protocol deviations or events that may affect the integrity of the PD data. Overall number of participants analyzed indicates the number of participants with data available for analyses. Number analyzed indicates the number of participants with data available for analyses in the specified category.
Measure: Mean (Standard Deviation); unit: percentage of VWF:Ag
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 23 | 21 | 19
percentage of VWF:Ag
  VWF:Ag : PK-I: number analyzed (Participants) | 23 | 0 | 19
  VWF:Ag : PK-I | -0.11 (17.064) |  | 3.67 (19.705)
  VWF:Ag : PK-II: number analyzed (Participants) | 22 | 21 | 0
  VWF:Ag : PK-II | 0.48 (34.798) | -1.31 (22.259) |
  VWF:Ag : PK-III: number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Assessment of Von Willebrand Factor:Ristocetin Cofactor Activity (VWF:RCo) During Prophylactic Treatment
Description: VWF:RCo provides a measure of the ability of VWF to bind platelet glycoprotein Ib. Stabilized platelets are agglutinated in the presence of VWF and the antibiotic Ristocetin. Assessments of VWF:RCo at baseline and following infusion of the SoC agent and TAK-755 treatment during the initial PK assessment was reported. PK-I, PK-II, and PK-III denote the crossover PK evaluation of a maximum of 14 days at the start of Prophylaxis Treatment Period 1 and end of Prophylaxis Treatment Periods 2 and 3 respectively. As per planned analysis, data for this outcome measure were collected and reported as per the treatment (intervention) received (rADAMTS13 manufactured in Orth, Austria [TAK-755 ORT], rADAMTS13 manufactured in Singapore [TAK-755 SIN], or SoC) during the course of the study, only for the prophylaxis cohorts. No participants received SoC in PK-II and PK-III thus there is no data for the same.
Time Frame: PK-I (Month 1:Day 12), PK-II (Month 12:Day 12), and PK-III (Month 19:Day 12): Post-infusion at 288 hours
Population: The PD Analysis Set included all FAS participants who had at least one valid data point for at least one of the PD outcome measures and had no major protocol deviations or events that may affect the integrity of the PD data. Overall number of participants analyzed indicates the number of participants with data available for analyses. Number analyzed indicates the number of participants with data available for analyses in the specified category.
Measure: Mean (Standard Deviation); unit: percentage of VWF:RCo
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 23 | 21 | 24
percentage of VWF:RCo
  VWF:RCo- PK-I: number analyzed (Participants) | 23 | 0 | 24
  VWF:RCo- PK-I | 3.63 (42.178) |  | 9.99 (33.230)
  VWF:RCo- PK-II: number analyzed (Participants) | 22 | 21 | 0
  VWF:RCo- PK-II | 7.45 (31.917) | 3.60 (30.678) |
  VWF:RCo- PK-III: number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Assessment of ADAMTS13 Activity Expressed as Pre-Infusion ADAMTS13 Levels
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Prophylaxis Cohort: TAK-755 ORT | Prophylaxis Cohort: TAK-755 SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 36 | 22 | 44
IU/mL
  ADAMTS13 Activity: PK-I: number analyzed (Participants) | 36 | 3 | 44
  ADAMTS13 Activity: PK-I | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification.
  ADAMTS13 Activity: PK-II: number analyzed (Participants) | 26 | 22 | 0
  ADAMTS13 Activity: PK-II | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. |
  ADAMTS13 Activity: PK-III: number analyzed (Participants) | 0 | 13 | 0
  ADAMTS13 Activity: PK-III |  | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. |

28. Secondary Outcome: Assessment of Select VWF Parameters Expressed as Pre-Infusion Levels of VWF:RCo
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of VWF:RCo
Groups:
- Prophylaxis Cohort: TAK-755-SIN: Participants received TAK-755 SIN dose of IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 SIN could also be given in Periods 1 and 2 depending on availability of TAK-755 ORT and other criteria.
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755-SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 36 | 25 | 43
percentage of VWF:RCo
  PK-I: VWF:RCo: number analyzed (Participants) | 36 | 5 | 43
  PK-I: VWF:RCo | 145.54 (54.698) | 137.62 (52.978) | 148.46 (51.415)
  PK-II: VWF:RCo: number analyzed (Participants) | 24 | 25 | 0
  PK-II: VWF:RCo | 155.76 (63.032) | 154.98 (74.444) |
  PK-III: VWF:RCo: number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Assessment of Select VWF Parameters Expressed as Pre-Infusion Levels of VWF:Ag
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of VWF:Ag
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755-SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 37 | 25 | 35
percentage of VWF:Ag
  PK-I: VWF:Ag: number analyzed (Participants) | 37 | 1 | 35
  PK-I: VWF:Ag | 110.38 (45.205) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 105.07 (40.539)
  PK-II: VWF:Ag: number analyzed (Participants) | 23 | 25 | 0
  PK-II: VWF:Ag | 120.48 (49.224) | 116.66 (60.338) |
  PK-III: VWF:Ag: number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Assessment of Select VWF Parameters Expressed as Pre-Infusion Levels of VWF:mm Low Resolution (Res.) Intermediate
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: % of VWF:mm Low Res.Intermediate
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755-SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 38 | 25 | 39
% of VWF:mm Low Res.Intermediate
  PK-I: VWF:mm Low Res. Intermediate: number analyzed (Participants) | 38 | 2 | 39
  PK-I: VWF:mm Low Res. Intermediate | 32.14 (3.375) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 31.22 (2.955)
  PK-II: VWF:mm Low Res. Intermediate: number analyzed (Participants) | 23 | 25 | 0
  PK-II: VWF:mm Low Res. Intermediate | 30.87 (3.754) | 31.10 (3.616) |
  PK-III: VWF:mm Low Res. Intermediate: number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Assessment of Select VWF Parameters Expressed as Pre-Infusion Levels of VWF:mm Low Res. Large
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: % of VWF:mm Low Res. Large
Groups:
- Prophylaxis Cohort: TAK-755-SIN: Participants received TAK-755 SIN prophylactic dose of IV infusions of 40 IU/kg Q2W for another 6 months in Period 3. TAK-755 SIN could also be given in Periods 1 and 2 depending on availability of TAK-755 ORT and other criteria.
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755-SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 38 | 25 | 39
% of VWF:mm Low Res. Large
  PK-I: VWF:mm Low Res. Large: number analyzed (Participants) | 38 | 2 | 39
  PK-I: VWF:mm Low Res. Large | 45.98 (5.920) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 46.03 (5.043)
  PK-II: VWF:mm Low Res. Large: number analyzed (Participants) | 23 | 25 | 0
  PK-II: VWF:mm Low Res. Large | 46.17 (5.670) | 44.93 (7.319) |
  PK-III: VWF:mm Low Res. Large: number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Assessment of Select VWF Parameters Expressed as Pre-Infusion Levels of VWF:mm Low Res. Small
Description: as for outcome 19
Time Frame: PK-I (Month 1:Day 1), PK-II (Month 12:Day 1), and PK-III (Month 19:Day 1): Pre-infusion (within 1 hour)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: % of VWF:mm Low Res. Small
Arm/Group | Prophylaxis Cohort: TAK-755-ORT | Prophylaxis Cohort: TAK-755-SIN | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 38 | 25 | 39
% of VWF:mm Low Res. Small
  PK-I: VWF:mm Low Res. Small: number analyzed (Participants) | 38 | 2 | 39
  PK-I: VWF:mm Low Res. Small | 21.66 (4.230) | NA (NA) — Mean and SD were not estimable as the values were below the lower limit of quantification. | 22.77 (5.161)
  PK-II: VWF:mm Low Res. Small: number analyzed (Participants) | 23 | 25 | 0
  PK-II: VWF:mm Low Res. Small | 22.96 (3.047) | 23.96 (5.320) |
  PK-III: VWF:mm Low Res. Small: number analyzed (Participants) | 0 | 0 | 0

33. Secondary Outcome: Number of Participants With Total Binding Antibodies to ADAMTS13 During Prophylactic Treatment
Description: Total binding antibodies to ADAMTS13 were measured by an ELISA-based assay, detecting total immunoglobulins (IgG, IgA, and IgM). As per planned analysis, data for this outcome measure were collected and reported per sequence (Prophylaxis Cohort I: TAK-755 Then SoC and Prophylaxis Cohort II: SoC Then TAK-755) for the prophylaxis cohorts only.
Time Frame: Up to 79.6 months
Population: The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization. 2 participants randomized to Prophylaxis Cohort I received actual treatment as per Prophylaxis Cohort II and are presented per actual treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755
Number analyzed (Participants) | 21 | 27
Participants | 0 | 2

34. Secondary Outcome: Number of Participants With Neutralizing Antibodies to ADAMTS13 During Prophylactic Treatment
Description: Neutralizing antibodies were measured by a Bethesda method with Nijmegen modification using the ADAMTS13 FRETS-VWF73 activity assay. As per planned analysis, data for this outcome measure were collected and reported per sequence (Prophylaxis Cohort I: TAK-755 Then SoC and Prophylaxis Cohort II: SoC Then TAK-755) for the prophylaxis cohorts only.
Time Frame: Up to 79.6 months
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755
Number analyzed (Participants) | 21 | 27
Participants | 0 | 1

35. Secondary Outcome: Number of Participants With Anti-Chinese Hamster Ovary (Anti-CHO) Protein Antibodies During Prophylactic Treatment
Description: Total immunoglobulin antibodies (Immunoglobulin G [IgG], A [IgA], and M [IgM]) against CHO protein were analyzed using ELISA assay. As per planned analysis, data for this outcome measure were collected and reported per sequence (Prophylaxis Cohort I: TAK-755 Then SoC and Prophylaxis Cohort II: SoC Then TAK-755) for the prophylaxis cohorts only.
Time Frame: Up to 79.6 months
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis Cohort I: TAK-755 Then SoC | Prophylaxis Cohort II: SoC Then TAK-755
Number analyzed (Participants) | 21 | 27
Participants | 0 | 2

36. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in cTTP-Patient Experience Questionnaire (cTTP-PEQ) Total Score
Description: The cTTP-PEQ consists of 26 questions designed to assess the participant's experience of fatigue, joint, muscle, abdominal &chest pain in the previous 24 hours, neurologic manifestations, bruising, feelings of depression and mood alterations, and activity limitation in the past 7 days, and participant's attitudes, experienced side effects, work/school absences and travel impact associated with treatment received for TTP during the previous 2 weeks. The cTTP PEQ is focused on measuring the symptoms and impacts of disease. The total scores range from 0 to 162. A higher score indicates greater burden and poor quality of life. As per planned analysis,for the prophylaxis cohorts the data for this outcome measure were collected and reported by categorizing as per Prophylaxis Periods and per age groups,≥12 years,12 to 18 years,≥18 years for both on demand(OD) and prophylaxis cohorts. No participants in the OD Cohorts had cTTP-PEQ data available for analysis at scheduled post-baseline visits.
Time Frame: Baseline, Urgent Treatment Period: Day 7, End of Period 1 (Month 6), End of Period 2 (Month 12), and End of Period 3 (Month 19)
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- On Demand Cohort I: TAK-755: Participants experiencing an acute TTP event who met all other inclusion criteria and entered the study through the TAK-755 cohort of the Urgent Treatment Period received initial dose of IV infusions 40 IU/kg [+/- 4 IU/kg] TAK-755 ORT or TAK-755 SIN infusion on Day 1 followed by a subsequent dose IV infusions of 20 IU/kg [+/- 2 IU/kg] TAK-755 ORT or TAK-755 SIN on Day 2 and an additional daily dose IV infusions of 15 IU/kg [+/- 1.5 IU/kg] TAK-755 on Day 3 until 2 days after the acute event was resolved. Upon resolution of the acute TTP event, participants had the option to either move to the prophylaxis cohort of the study or discontinue entirely.
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 22 | 12 | 0 | 0
score on a scale
  ≥12 years: Total Score, Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  ≥12 years: Total Score, End of Period 1: number analyzed (Participants) | 9 | 12 | 0 | 0
  ≥12 years: Total Score, End of Period 1 | -2.6 (24.17) | -2.2 (12.47) |  |
  ≥12 years: Total Score, End of Period 2: number analyzed (Participants) | 12 | 8 | 0 | 0
  ≥12 years: Total Score, End of Period 2 | -10.4 (18.13) | -1.4 (18.38) |  |
  ≥12 years: Total Score, End of Period 3: number analyzed (Participants) | 22 | 0 | 0 | 0
  ≥12 years: Total Score, End of Period 3 | -10.6 (13.13) |  |  |
  12 to < 18 years: Total Score, Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  12 to < 18 years: Total Score, End of Period 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  12 to < 18 years: Total Score, End of Period 1 |  | 12.0 (NA) — SD was not estimable for a single participant. |  |
  12 to < 18 years: Total Score, End of Period 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  12 to < 18 years: Total Score, End of Period 2 | 13.0 (NA) — SD was not estimable for a single participant. |  |  |
  12 to < 18 years: Total Score, End of Period 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  12 to < 18 years: Total Score, End of Period 3 | -6.0 (NA) — SD was not estimable for a single participant. |  |  |
  ≥18 years: Total Score, Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  ≥18 years: Total Score, End of Period 1: number analyzed (Participants) | 9 | 11 | 0 | 0
  ≥18 years: Total Score, End of Period 1 | -2.6 (24.17) | -3.5 (12.22) |  |
  ≥18 years: Total Score, End of Period 2: number analyzed (Participants) | 11 | 8 | 0 | 0
  ≥18 years: Total Score, End of Period 2 | -12.5 (17.37) | -1.4 (18.38) |  |
  ≥18 years: Total Score, End of Period 3: number analyzed (Participants) | 21 | 0 | 0 | 0
  ≥18 years: Total Score, End of Period 3 | -10.9 (13.41) |  |  |

37. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in Physical and Mental Component Scores of the 36-Item Short Form Health Survey Version 2 (SF-36v2)
Description: SF-36v2 is questionnaire that evaluated participant's health related quality of life. It included 36 questions related to 8 health dimensions: physical functioning, role-physical(role limitations due to physical health problems), bodily pain, general health, vitality(energy/fatigue),social functioning, role-emotional(role limitations due to emotional problems),& mental health. Based on these 4 scales(physical functioning, role-physical, bodily pain, general health), physical component score was generated which ranges between 0 &100, with higher scores indicating a better quality of life. Based on these 4 scales(vitality, social functioning, role-emotional,&mental health), mental component score was generated ranging between 0&100, with higher scores=better quality of life. As per planned analysis, for the prophylaxis cohorts data for this outcome measure were collected&reported by categorizing as per Prophylaxis Periods and per component scores for both on demand&prophylaxis cohorts.
Time Frame: as for outcome 36
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category. No participants in the OD Cohorts had SF-36v2 data available for analysis at scheduled post-baseline visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 21 | 11 | 0 | 0
score on a scale
  Physical Component Score: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Physical Component Score: End of Period 1: number analyzed (Participants) | 9 | 11 | 0 | 0
  Physical Component Score: End of Period 1 | 3.934 (10.1098) | -0.532 (4.8297) |  |
  Physical Component Score: End of Period 2: number analyzed (Participants) | 12 | 8 | 0 | 0
  Physical Component Score: End of Period 2 | 3.121 (6.3196) | 2.625 (6.4219) |  |
  Physical Component Score: End of Period 3: number analyzed (Participants) | 21 | 0 | 0 | 0
  Physical Component Score: End of Period 3 | 1.019 (4.8970) |  |  |
  Mental Component Score: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Mental Component Score: End of Period 1: number analyzed (Participants) | 9 | 11 | 0 | 0
  Mental Component Score: End of Period 1 | -7.263 (7.4244) | 5.418 (5.0244) |  |
  Mental Component Score: End of Period 2: number analyzed (Participants) | 12 | 8 | 0 | 0
  Mental Component Score: End of Period 2 | 2.880 (5.2646) | -4.853 (9.9302) |  |
  Mental Component Score: End of Period 3: number analyzed (Participants) | 21 | 0 | 0 | 0
  Mental Component Score: End of Period 3 | 3.852 (7.4066) |  |  |

38. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in Abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) Domain Scores
Description: TSQM is a treatment satisfaction measure used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are treatment effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicates greater satisfaction in that domain. As per planned analysis, for the prophylaxis cohorts data for this outcome measure were collected and reported by categorizing as per Prophylaxis Periods and per domain scores for both on demand and prophylaxis cohorts.
Time Frame: as for outcome 36
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category. No participants in the OD Cohorts had TSQM-9 data available for analysis at scheduled post-baseline visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 19 | 10 | 0 | 0
score on a scale
  Treatment Effectiveness Score: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Treatment Effectiveness Score: End of Period 1: number analyzed (Participants) | 6 | 10 | 0 | 0
  Treatment Effectiveness Score: End of Period 1 | 26.8519 (36.07548) | 4.4444 (13.55778) |  |
  Treatment Effectiveness Score: End of Period 2: number analyzed (Participants) | 10 | 6 | 0 | 0
  Treatment Effectiveness Score: End of Period 2 | 25.0000 (17.42119) | 12.9630 (17.09330) |  |
  Treatment Effectiveness Score: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Treatment Effectiveness Score: End of Period 3 | 22.2222 (20.11626) |  |  |
  Convenience Score: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Convenience Score: End of Period 1: number analyzed (Participants) | 6 | 10 | 0 | 0
  Convenience Score: End of Period 1 | 36.1111 (16.75900) | 1.6667 (11.43059) |  |
  Convenience Score: End of Period 2: number analyzed (Participants) | 10 | 6 | 0 | 0
  Convenience Score: End of Period 2 | 27.7778 (15.27076) | 14.8148 (27.81479) |  |
  Convenience Score: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Convenience Score: End of Period 3 | 21.0526 (29.48919) |  |  |
  Global Satisfaction Score: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Global Satisfaction Score: End of Period 1: number analyzed (Participants) | 6 | 10 | 0 | 0
  Global Satisfaction Score: End of Period 1 | 28.5714 (9.03508) | 5.0000 (16.85270) |  |
  Global Satisfaction Score: End of Period 2: number analyzed (Participants) | 10 | 6 | 0 | 0
  Global Satisfaction Score: End of Period 2 | 23.5714 (16.85270) | 14.2857 (21.66536) |  |
  Global Satisfaction Score: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Global Satisfaction Score: End of Period 3 | 22.9323 (16.07433) |  |  |

39. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in EuroQoL 5 Dimensions Questionnaire 3-Level (EQ-5D-3L) Domain Scores
Description: EQ-5D-3L health questionnaire is a participant-answered questionnaire scoring 5 dimensions(domains) - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on an ordinal scale with 3 available levels of response and scores ranging from 1 to 3, "no problems," "some problems," and "extreme problems," respectively. Lower scores for the domains in the EQ-5D-3L indicate improvement. As per planned analysis, for the prophylaxis cohorts data for this outcome measure were collected and reported by categorizing as per Prophylaxis Periods and per domain scores for both on demand and prophylaxis cohorts.
Time Frame: as for outcome 36
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category. No participants in the OD Cohorts had EQ-5D-3L data available for analysis at scheduled post-baseline visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 19 | 10 | 0 | 0
score on a scale
  Mobility: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Mobility: End of Period 1: number analyzed (Participants) | 8 | 10 | 0 | 0
  Mobility: End of Period 1 | 0.3 (0.46) | -0.1 (0.32) |  |
  Mobility: End of Period 2: number analyzed (Participants) | 11 | 6 | 0 | 0
  Mobility: End of Period 2 | -0.1 (0.30) | 0.0 (0.00) |  |
  Mobility: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Mobility: End of Period 3 | -0.1 (0.23) |  |  |
  Self-Care: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Self-Care: End of Period 1: number analyzed (Participants) | 8 | 10 | 0 | 0
  Self-Care: End of Period 1 | 0.1 (0.35) | 0.0 (0.00) |  |
  Self-Care: End of Period 2: number analyzed (Participants) | 11 | 6 | 0 | 0
  Self-Care: End of Period 2 | 0.0 (0.00) | 0.0 (0.00) |  |
  Self-Care: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Self-Care: End of Period 3 | -0.1 (0.23) |  |  |
  Usual Activities: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Usual Activities: End of Period 1: number analyzed (Participants) | 8 | 10 | 0 | 0
  Usual Activities: End of Period 1 | 0.0 (0.53) | -0.2 (0.42) |  |
  Usual Activities: End of Period 2: number analyzed (Participants) | 11 | 6 | 0 | 0
  Usual Activities: End of Period 2 | 0.0 (0.45) | 0.0 (0.63) |  |
  Usual Activities: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Usual Activities: End of Period 3 | -0.1 (0.40) |  |  |
  Pain/Discomfort: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Pain/Discomfort: End of Period 1: number analyzed (Participants) | 8 | 10 | 0 | 0
  Pain/Discomfort: End of Period 1 | 0.3 (0.46) | -0.2 (0.63) |  |
  Pain/Discomfort: End of Period 2: number analyzed (Participants) | 11 | 6 | 0 | 0
  Pain/Discomfort: End of Period 2 | -0.3 (0.65) | 0.2 (0.41) |  |
  Pain/Discomfort: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Pain/Discomfort: End of Period 3 | -0.2 (0.54) |  |  |
  Anxiety/Depression: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Anxiety/Depression: End of Period 1: number analyzed (Participants) | 8 | 10 | 0 | 0
  Anxiety/Depression: End of Period 1 | 0.1 (0.64) | 0.0 (0.00) |  |
  Anxiety/Depression: End of Period 2: number analyzed (Participants) | 11 | 6 | 0 | 0
  Anxiety/Depression: End of Period 2 | -0.1 (0.30) | 0.0 (0.00) |  |
  Anxiety/Depression: End of Period 3: number analyzed (Participants) | 19 | 0 | 0 | 0
  Anxiety/Depression: End of Period 3 | -0.1 (0.46) |  |  |

40. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in EQ-5D-youth (EQ-5D-Y) Domain Scores
Description: EQ-5D-Y health questionnaire is a participant answered questionnaire scoring 5 dimensions (domains) - mobility, self-care, usual activities, pain/discomfort and anxiety/depression assessed in participants aged from 8 to 16 years. The EQ-5D-Y descriptive system includes 5 descriptive items: Mobility, self-care, doing usual activities, having pain or discomfort, and feeling anxiety or depressed. Each dimension is scored at 3 levels: 1=No problems, 2=some problems, and 3=a lot of problems. Lower scores for the domains in the EQ-5D-Y indicate improvement. As per planned analysis, for the prophylaxis cohorts data for this outcome measure were collected and reported by categorizing as per Prophylaxis Periods and per domain scores for both on demand and prophylaxis cohorts.
Time Frame: as for outcome 36
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category. No participants in the OD Cohorts had EQ-5D-Y data available for analysis at scheduled post-baseline visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 4 | 3 | 0 | 0
score on a scale
  Mobility: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Mobility: End of Period 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Mobility: End of Period 1 | 0.0 (NA) — SD was not estimable for a single participant. | 0.0 (0.00) |  |
  Mobility: End of Period 2: number analyzed (Participants) | 3 | 1 | 0 | 0
  Mobility: End of Period 2 | 0.0 (0.00) | 0.0 (NA) — SD was not estimable for a single participant. |  |
  Mobility: End of Period 3: number analyzed (Participants) | 4 | 0 | 0 | 0
  Mobility: End of Period 3 | 0.0 (0.00) |  |  |
  Self-Care: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Self-Care: End of Period 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Self-Care: End of Period 1 | 0.0 (NA) — SD was not estimable for a single participant. | 0.0 (0.00) |  |
  Self-Care: End of Period 2: number analyzed (Participants) | 3 | 1 | 0 | 0
  Self-Care: End of Period 2 | 0.0 (0.00) | 0.0 (NA) — SD was not estimable for a single participant. |  |
  Self-Care: End of Period 3: number analyzed (Participants) | 4 | 0 | 0 | 0
  Self-Care: End of Period 3 | 0.0 (0.00) |  |  |
  Usual Activities: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Usual Activities: End of Period 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Usual Activities: End of Period 1 | 0.0 (NA) — SD was not estimable for a single participant. | 0.0 (0.00) |  |
  Usual Activities: End of Period 2: number analyzed (Participants) | 3 | 1 | 0 | 0
  Usual Activities: End of Period 2 | 0.0 (0.00) | 0.0 (NA) — SD was not estimable for a single participant. |  |
  Usual Activities: End of Period 3: number analyzed (Participants) | 4 | 0 | 0 | 0
  Usual Activities: End of Period 3 | 0.0 (0.00) |  |  |
  Pain/Discomfort: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Pain/Discomfort: End of Period 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Pain/Discomfort: End of Period 1 | 1.0 (NA) — SD was not estimable for a single participant. | -0.7 (0.58) |  |
  Pain/Discomfort: End of Period 2: number analyzed (Participants) | 3 | 1 | 0 | 0
  Pain/Discomfort: End of Period 2 | -0.7 (0.58) | 0.0 (NA) — SD was not estimable for a single participant. |  |
  Pain/Discomfort: End of Period 3: number analyzed (Participants) | 4 | 0 | 0 | 0
  Pain/Discomfort: End of Period 3 | -0.3 (0.96) |  |  |
  Anxiety/Depression: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  Anxiety/Depression: End of Period 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Anxiety/Depression: End of Period 1 | 0.0 (NA) — SD was not estimable for a single participant. | 0.0 (0.00) |  |
  Anxiety/Depression: End of Period 2: number analyzed (Participants) | 3 | 1 | 0 | 0
  Anxiety/Depression: End of Period 2 | 0.3 (0.58) | 0.0 (NA) — SD was not estimable for a single participant. |  |
  Anxiety/Depression: End of Period 3: number analyzed (Participants) | 4 | 0 | 0 | 0
  Anxiety/Depression: End of Period 3 | 0.0 (0.00) |  |  |

41. Secondary Outcome: Health Related Quality of Life (HRQoL) Assessed as Change From Baseline in Pediatric Quality of Life Inventory (Peds QL) Scale Total Scores
Description: The PedsQL is a generic health related quality of life instrument designed specifically for a pediatric population and captures following domains: physical functioning, emotional functioning, social functioning, school functioning, psychosocial summary, physical health and total score. The Peds-QL total score consists of all 23 items of all domains. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better quality of life. As per planned analysis, for the prophylaxis cohorts data for this outcome measure were collected and reported by categorizing as per Prophylaxis Periods and per age groups, 2 to < 5 years, 5 to < 8 years, 8 to < 13 years, and 13 to < 18 years, for both on demand and prophylaxis cohorts.
Time Frame: as for outcome 36
Population: Modified FAS. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for specified category. No participants in the OD Cohorts had Peds QL data available for analysis at scheduled post-baseline visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
Number analyzed (Participants) | 7 | 5 | 0 | 0
score on a scale
  2 to < 5 years: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  2 to < 5 years, End of Period 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  2 to < 5 years, End of Period 1 | 25.0000 (47.14045) |  |  |
  2 to < 5 years, End of Period 2: number analyzed (Participants) | 0 | 2 | 0 | 0
  2 to < 5 years, End of Period 2 |  | 27.3810 (47.14045) |  |
  2 to < 5 years, End of Period 3: number analyzed (Participants) | 2 | 0 | 0 | 0
  2 to < 5 years, End of Period 3 | 24.4048 (49.66583) |  |  |
  5 to < 8 years: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  5 to < 8 years, End of Period 1: number analyzed (Participants) | 1 | 1 | 0 | 0
  5 to < 8 years, End of Period 1 | 29.3478 (NA) — SD was not estimable for a single participant. | -16.3043 (NA) — SD was not estimable for a single participant. |  |
  5 to < 8 years, End of Period 2: number analyzed (Participants) | 1 | 1 | 0 | 0
  5 to < 8 years, End of Period 2 | -6.5217 (NA) — SD was not estimable for a single participant. | 32.6087 (NA) — SD was not estimable for a single participant. |  |
  5 to < 8 years, End of Period 3: number analyzed (Participants) | 2 | 0 | 0 | 0
  5 to < 8 years, End of Period 3 | 17.9348 (19.21486) |  |  |
  8 to < 13 years: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  8 to < 13 years, End of Period 1: number analyzed (Participants) | 1 | 2 | 0 | 0
  8 to < 13 years, End of Period 1 | -2.1739 (NA) — SD was not estimable for a single participant. | 15.2174 (13.83470) |  |
  8 to < 13 years, End of Period 2: number analyzed (Participants) | 2 | 1 | 0 | 0
  8 to < 13 years, End of Period 2 | 8.6957 (23.05783) | 1.0870 (NA) — SD was not estimable for a single participant. |  |
  8 to < 13 years, End of Period 3: number analyzed (Participants) | 3 | 0 | 0 | 0
  8 to < 13 years, End of Period 3 | 5.7971 (7.39876) |  |  |
  13 to < 18 years: Urgent Treatment Period Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0
  13 to < 18 years, End of Period 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  13 to < 18 years, End of Period 2: number analyzed (Participants) | 0 | 0 | 0 | 0
  13 to < 18 years, End of Period 3: number analyzed (Participants) | 0 | 0 | 0 | 0

42. Secondary Outcome: Resource Utilization: Annualized Length of Hospital Stay for Acute TTP Events for Prophylaxis Cohorts
Description: The annualized number of days participants stayed in hospital for acute TTP events were assessed. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts in a combined manner for Periods 1 and 2 for SoC treatment and for Periods 1, 2, and 3 for TAK-755 treatment respectively.
Time Frame: Up to 79.6 months
Population: Modified FAS included all FAS participants who were treated according to their randomized treatment sequence with the exclusion of those enrolled prior to November 2017 who were treated with SoC instead of the randomized treatment of TAK-755 in period 1 because TAK-755 was not available. For participants enrolled prior to November 2017, only the first 6 months of SoC treatment in period 1 was included in the analysis.
Measure: Median (Full Range); unit: days/year
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 44 | 45
days/year | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 3.4]

43. Secondary Outcome: Resource Utilization: Annualized Number of Acute Care Visits for Prophylaxis Cohorts
Description: Annualized number of acute care visits was calculated as the number of acute care visits × 365.25/(End date - treatment start date + 1). As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts in a combined manner for Periods 1 and 2 for SoC treatment and for Periods 1, 2, and 3 for TAK-755 treatment respectively.
Time Frame: Up to 79.6 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: acute care visits per year
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 44 | 45
acute care visits per year | 0.60 (1.331) | 0.14 (0.498)

44. Secondary Outcome: Resource Utilization: Annualized Number of Days Missed From School or Work for Prophylaxis Cohorts
Description: Annualized number of days missed from school or work were assessed. As per planned analysis, data for this outcome measure were collected and reported only for the prophylaxis cohorts in a combined manner for Periods 1 and 2 for SoC treatment and for Periods 1, 2, and 3 for TAK-755 treatment respectively.
Time Frame: Up to 79.6 months
Population: as for outcome 42
Measure: Median (Full Range); unit: days/year
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC
Number analyzed (Participants) | 44 | 45
days/year | 0.00 [0.0 to 180.3] | 0.00 [0.0 to 294.5]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (79.6 months)
Description: The Safety Analysis Set included all participants treated with at least 1 dose of TAK-755 or SoC treatment after randomization. As per planned analysis, data for adverse events were collected and reported in a combined manner irrespective of the Prophylaxis Periods and partitioned as per the treatment received during the course of the study, presented for the on demand and prophylaxis cohorts.
Arm/Group | Prophylaxis Cohort: TAK-755 | Prophylaxis Cohort: SoC | On Demand Cohort I: TAK-755 | On Demand Cohort II: SoC
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 6/47 | 8/48 | 0/2 | 1/4
Other Adverse Events (participants affected / at risk) | 39/47 | 37/48 | 0/2 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis Cohort: TAK-755 (N=47) | Prophylaxis Cohort: SoC (N=48) | On Demand Cohort I: TAK-755 (N=2) | On Demand Cohort II: SoC (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis Cohort: TAK-755 (N=47) | Prophylaxis Cohort: SoC (N=48) | On Demand Cohort I: TAK-755 (N=2) | On Demand Cohort II: SoC (N=4)
Abdominal pain (Gastrointestinal disorders) | 8 | 6 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 7 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0
Asthenia (General disorders) | 3 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 8 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0
Fatigue (General disorders) | 5 | 7 | 0 | 0
Haematoma (Vascular disorders) | 3 | 2 | 0 | 0
Headache (Nervous system disorders) | 15 | 10 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Lethargy (Nervous system disorders) | 5 | 3 | 0 | 0
Malaise (General disorders) | 3 | 2 | 0 | 0
Migraine (Nervous system disorders) | 7 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 2 | 0 | 1
Oral herpes (Infections and infestations) | 3 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 0 | 0 | 0
Platelet count decreased (Investigations) | 4 | 5 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1
Pyrexia (General disorders) | 6 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0
Rhinitis (Infections and infestations) | 7 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 3 | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 7 | 0 | 0
Viral infection (Infections and infestations) | 4 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 6 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03393975/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT03393975/SAP_001.pdf